CLINICAL TRIAL: NCT01135290
Title: Evaluation of HP828-101 for Post Treatment Care Following a Chemical Peel or Laser Resurfacing
Brief Title: Post Treatment Care After Chemical Peel or Laser Resurfacing
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Business decision, formulation will not be pursued.
Sponsor: Healthpoint (Industry)
Responsible Party: Herbert B. Slade, MD FAAAAI / Chief Medical Officer, Healthpoint, Ltd
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 828-101-09-016
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Chemical Peel
Keywords: The management of post-treatment symptoms for subjects that had either a medium grade chemical peel or fractional resurfacing
MeSH Terms: interventions — Petrolatum

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Other)
  Interventions: Drug: Aquaphor
- A (Active Comparator)
  Interventions: Drug: HP828-101

INTERVENTIONS:
Drug: Aquaphor
  Arms: B
Drug: HP828-101
  Arms: A

SUMMARY:
This study tests two different approaches to the resolution of facial skin resurfacing.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent document and photography release must be read, signed, and dated by the subject or the subject's legally authorized representative before conducting any study procedures or exams. In addition, the informed consent and photography release document must be signed and dated by the individual who consents the subject before conducting Visit 1. A photocopy of the signed informed consent document must be provided to the subject, and the original signed document placed in the subject's chart.
* Subjects 18 years of age or older, scheduled to undergo either a medium chemical peel with 35% TCA or a laser resurfacing. Subjects may be of either sex and of any race or skin type provided that their skin color, in the opinion of the Investigator, will not interfere with the study assessments.
* Women of child-bearing potential (those who are not premenarchal, not surgically sterilized [hysterectomy or bilateral oophorectomy], or not post-menopausal) may participate in the study if they meet all of the following conditions:

  * they are not breast feeding
  * undertake a pregnancy test, which must be negative
  * they do not intend to become pregnant during the study
  * they are using adequate birth control methods and they agree to continue using those methods for the duration of the study

Adequate birth control methods are defined as: hormonal-topical, oral, implantable, or injectable contraceptives; mechanical-spermicide in conjunction with a barrier such as a condom or diaphragm; IUD; or, surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use an adequate birth control method as described above for the remainder of the study.

NOTE: Women who have had a bilateral tubal ligation are not considered to have been surgically sterilized and must agree to the conditions as specified above.

* Willing and able to make all required study visits.
* Able to follow instructions.
* Undergo a medium grade chemical peel or fractional resurfacing.

Exclusion Criteria:

* Contraindications or hypersensitivity to the use of the study medications or their components (e.g., balsam of Peru, castor oil, or phenoxyethanol).
* Therapy with another investigational agent within thirty (30) days of Visit 1, or during the study.
* Have taken anticoagulants (blood thinners, including aspirin) within two weeks.
* Current smoker.
* Use of oral isotretinoin during the past 12 months, systemic steroids, topical retinoids, or topical corticosteroids within the month prior to the study.
* Have any congenital skin disorder which affects keratinocytes, elastin, or collagen.
* Have any dermatologic disease which may be aggravated or provoked by the wounding procedure.
* Are at risk of keloid or hypertrophic scar formation based on personal or family history, or skin exam.
* Have any skin disorder which causes delayed healing.
* Have any systemic condition that would compromise skin healing.
* The Medical Monitor may declare any subject ineligible for a valid medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Physician and subject evaluation ratings of the signs and symptoms of facial skin during post-operative care. | 84 Days

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Jeffery Kenkel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States